CLINICAL TRIAL: NCT05273632
Title: Comparison Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate Versus Placebo to Reduce Blood Loss Intraoperative and Post Operative During Elective Cesarean Section
Brief Title: Comparison Study of Oxytocin Versus Tranexamic Acid and Etamsylaye Versus Placebo(Saline)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EL-SAYED EL-DESOUKY
Record Dates: First submitted 2020-12-02; First posted 2022-03-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Blood Loss, Surgical; Blood Loss, Postoperative
Keywords: blood loss; cesarean section; oxytocin; tranexamic acid; etamsylate; saline; Intra-operative; Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage; Hemorrhage | interventions — Oxytocin; Tranexamic Acid; Ethamsylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin (Active Comparator): Pre- Operative Oxytocin is given intravenously 5-10 minutes slowly before skin incision
  Interventions: Drug: Oxytocin
- Tranexamic acid and Etamsylate (Active Comparator): Tranexamic acid and Etamsylate are slowly given intravenously 10 minutes before start of Cesarean Delivery
  Interventions: Drug: Oxytocin
- Saline (Placebo Comparator): Normal saline (about 200 ml) is given intravenously 10 minutes before start of Cesarean Section
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — trial of reduction of losing blood intra operative or post operative during Cesarean Delivery
  Other Names: Tranexamic acid and Etamsylate

SUMMARY:
Comparison Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate Versus Normal Saline as Pre-operative Administration.

DETAILED DESCRIPTION:
Comparison Study Between Oxytocin Versus Tranexamic Acid and Ethamsylate Versus Normal Saline to reduce intra operative bleeding and postoperative bleeding during elective Cesarean Delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females admitted for Elective Cesarean Section.
* Gestational age of pregnancy (38 weeks To 40 weeks).
* the average height of 145 to 160 cm,average body weight of 45 to 85 kgs.
* Singleton living fetus.
* No medical disorders.
* Informed Oral Consent From The Patient.

Exclusion Criteria:

* Severe medical and surgical disorders as thyroid dysfunction, which was excluded by routine thyroid function test (free T3, free T4, and thyroid stimulating hormone(TSH), all of them should be within normal limits).
* Bleeding tendency, for example, disseminated intravascular coagulopathy, which was excluded by platelet count, coagulation time, bleeding time, prothrombin time, partial thromboplastin time, and thrombin time (all should be within normal).
* Acute liver or kidney diseases; blood disorders, such as anaemia.
* Allergy to Tranexamic acid.
* Risk factors for PPH, such as polyhydramnios, fetal macrosomia, antepartum haemorrhage.
* Ante partum Hemorrhage such placental abruption.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
blood loss during and after cesarean delivery | First 2 hours after C-Section
  Measuring of Hemoglobin level and Hematocrit level pre and post operatively.

SECONDARY OUTCOMES:
post operative bleeding | first 24 hours after C-Section
  assessment of Hemoglobin level and Hematocrit level post operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sayed Galal Hospital, Alhusein Hospital, Alzahraa Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No